CLINICAL TRIAL: NCT00474435
Title: The Pharmacokinetics of Co-formulated Emtricitabine/Tenofovir/Efavirenz in HIV-infected Patients With Smear-positive Pulmonary Tuberculosis in the Kilimanjaro Region, Tanzania
Brief Title: Pharmacokinetics of Emtricitabine/Tenofovir/Efavirenz in HIV-infected Patients With Tuberculosis
Acronym: PETE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: African Poverty Related Infection Oriented Research Initiative (Other)
Collaborators: Radboud University Medical Center (Other); Kilimanjaro Christian Medical Centre, Tanzania (Other)
Responsible Party: Martin Boeree, University Lungcentre Dekkerswald, Groesbeek, the Netherlands
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCN-AKF 04.03
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2008-12

CONDITIONS: Tuberculosis; HIV Infections
Keywords: Tuberculosis; HIV; Coinfection; Pharmacokinetics; Emtricitabine; Tenofovir; Rifampin; Efavirenz; Treatment Naive
MeSH Terms: conditions — Tuberculosis; HIV Infections; Coinfection | interventions — Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Emtricitabine/tenofovir/efavirenz — Co-formulated in one tablet (taken once daily by oral administration):
  * emtricitabine 200 mg
  * tenofovir DF 300 mg
  * efavirenz 600 mg

SUMMARY:
In this pilot study the pharmacokinetics and safety of the antiretroviral combination of co-formulated emtricitabine/tenofovir/efavirenz will be studied in HIV-positive patients with pulmonary tuberculosis (TB) who are concomitantly treated with a standard rifampin-containing tuberculostatic regimen. It is expected that this antiretroviral combination causes minimal drug interactions with the rifampin-containing anti-tuberculosis medication.

DETAILED DESCRIPTION:
The primary objectives of this pilot study in 30 patients are:

1. To determine the effect of rifampin-containing tuberculostatic treatment on the pharmacokinetic profile of emtricitabine+tenofovir+efavirenz, when co-formulated in one tablet, in HIV-infected patients with smear-positive pulmonary tuberculosis in Tanzania.
2. To determine the effect of the emtricitabine+tenofovir+efavirenz regimen on the pharmacokinetics of tuberculostatics in the same population.

The secondary objectives are:

1. To determine the safety of co-administration of emtricitabine+tenofovir+efavirenz with treatment for smear-positive pulmonary tuberculosis.
2. To determine the short-term (24 weeks) virological efficacy on HIV of an emtricitabine+tenofovir+efavirenz regimen in patients with smear-positive pulmonary tuberculosis.
3. To determine the short-term bacteriological efficacy on smear-positive tuberculosis of the co-administration of a standard regimen for tuberculosis and an emtricitabine+tenofovir+efavirenz regimen.

ELIGIBILITY:
Inclusion Criteria:

* A smear-positive pulmonary tuberculosis, based on positive smear of at least two sputum samples with Ziehl-Neelsen (ZN) staining.
* HIV-infected as documented by positive HIV antibody test.
* Subject is at least 18 years of age at the day of the first dosing of study medication.
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
* CD4 cell count > 50 copies/mm3.
* Karnofsky score > 40.
* Willing and able to regularly attend the Kibung'oto National Tuberculosis Hospital (KNTH) clinic.

Exclusion Criteria:

* History of sensitivity/idiosyncrasy to the drug or chemically related compounds or excipients, which may be employed in the trial.
* Previously treated for HIV infection with antiretroviral agents.
* Pregnant or breastfeeding.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* A history of severe psychiatric disease such as psychosis, schizophrenia, etc.
* Inability to understand the nature and extent of the trial and the procedures required.
* Abnormal serum transaminases or creatinine, determined as levels being > 5 times upper limit of normal.
* Active hepatobiliary or hepatic disease (Non B Chronic Hepatitis B/C co-infection is allowed).
* CD4 cell count > 350 cells/mm3.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of emtricitabine, tenofovir and efavirenz | Two 24 hour pharmacokinetic (PK) curves (week 8 and 28)
Pharmacokinetic parameters of the tuberculostatic agents | Pharmacokinetic (PK) samples at 2 hours and 6 hours postdose (week 2 and 8)

SECONDARY OUTCOMES:
Biochemistry and haematology samples for safety | Samples at screening, baseline, week 2, 4, 6, 8, 12, 16, 24, 28
Questioning about occurrence of adverse events | At baseline, week 2, 4, 6, 8, 12, 16, 24, 28
CD4 count and HIV-1 RNA | At screening, week 4, week 16 and week 28
Sputum staining and culture | At screening, week 4, 8, and 28

CONTACTS AND LOCATIONS:
Overall Officials: Martin Boeree, MD, PhD, Principal Investigator — University Lungcentre Dekkerswald, Groesbeek / University Medical Centre Nijmegen, the Netherlands; David Burger, PharmD, PhD, Principal Investigator — University Medical Centre Nijmegen, the Netherlands; Gibson Kibiki, MMed, PhD, Principal Investigator — Kilimanjaro Christian Medical Centre,Moshi,Tanzania
Locations (1):
- Kibong'oto National Tuberculosis Hospital, Moshi, Kilimanjaro, Tanzania

REFERENCES:
- [Background] Bowen EF, Rice PS, Cooke NT, Whitfield RJ, Rayner CF. HIV seroprevalence by anonymous testing in patients with Mycobacterium tuberculosis and in tuberculosis contacts. Lancet. 2000 Oct 28;356(9240):1488-9. doi: 10.1016/S0140-6736(00)02876-2. PMID 11081535
- [Background] Msamanga GI, Fawzi WW. The double burden of HIV infection and tuberculosis in sub-Saharan Africa. N Engl J Med. 1997 Sep 18;337(12):849-51. doi: 10.1056/NEJM199709183371210. No abstract available. PMID 9295244
- [Background] Dean GL, Edwards SG, Ives NJ, Matthews G, Fox EF, Navaratne L, Fisher M, Taylor GP, Miller R, Taylor CB, de Ruiter A, Pozniak AL. Treatment of tuberculosis in HIV-infected persons in the era of highly active antiretroviral therapy. AIDS. 2002 Jan 4;16(1):75-83. doi: 10.1097/00002030-200201040-00010. PMID 11741165
- [Background] Burman WJ, Gallicano K, Peloquin C. Comparative pharmacokinetics and pharmacodynamics of the rifamycin antibacterials. Clin Pharmacokinet. 2001;40(5):327-41. doi: 10.2165/00003088-200140050-00002. PMID 11432536
- [Background] Finch CK, Chrisman CR, Baciewicz AM, Self TH. Rifampin and rifabutin drug interactions: an update. Arch Intern Med. 2002 May 13;162(9):985-92. doi: 10.1001/archinte.162.9.985. PMID 11996607
- [Background] Lopez-Cortes LF, Ruiz-Valderas R, Viciana P, Alarcon-Gonzalez A, Gomez-Mateos J, Leon-Jimenez E, Sarasanacenta M, Lopez-Pua Y, Pachon J. Pharmacokinetic interactions between efavirenz and rifampicin in HIV-infected patients with tuberculosis. Clin Pharmacokinet. 2002;41(9):681-90. doi: 10.2165/00003088-200241090-00004. PMID 12126459
- [Background] Burger DM, Meenhorst PL, Koks CH, Beijnen JH. Pharmacokinetic interaction between rifampin and zidovudine. Antimicrob Agents Chemother. 1993 Jul;37(7):1426-31. doi: 10.1128/AAC.37.7.1426. PMID 8363370
- [Background] Gallicano KD, Sahai J, Shukla VK, Seguin I, Pakuts A, Kwok D, Foster BC, Cameron DW. Induction of zidovudine glucuronidation and amination pathways by rifampicin in HIV-infected patients. Br J Clin Pharmacol. 1999 Aug;48(2):168-79. doi: 10.1046/j.1365-2125.1999.00987.x. PMID 10417493
- [Background] Friedland G, Abdool Karim S, Abdool Karim Q, Lalloo U, Jack C, Gandhi N, El Sadr W. Utility of tuberculosis directly observed therapy programs as sites for access to and provision of antiretroviral therapy in resource-limited countries. Clin Infect Dis. 2004 Jun 1;38 Suppl 5:S421-8. doi: 10.1086/421407. PMID 15156433
- [Background] Droste JA, Aarnoutse RE, Koopmans PP, Hekster YA, Burger DM. Evaluation of antiretroviral drug measurements by an interlaboratory quality control program. J Acquir Immune Defic Syndr. 2003 Mar 1;32(3):287-91. doi: 10.1097/00126334-200303010-00007. PMID 12626888
- [Background] Holland DT, DiFrancesco R, Stone J, Hamzeh F, Connor JD, Morse GD; Adult and Pediatric AIDS Clinical Trials Group Pharmacology Laboratory Committees, Pediatric AIDS Clinical Trials Group. Quality assurance program for clinical measurement of antiretrovirals: AIDS clinical trials group proficiency testing program for pediatric and adult pharmacology laboratories. Antimicrob Agents Chemother. 2004 Mar;48(3):824-31. doi: 10.1128/AAC.48.3.824-831.2004. PMID 14982771
- [Background] Marzolini C, Telenti A, Decosterd LA, Greub G, Biollaz J, Buclin T. Efavirenz plasma levels can predict treatment failure and central nervous system side effects in HIV-1-infected patients. AIDS. 2001 Jan 5;15(1):71-5. doi: 10.1097/00002030-200101050-00011. PMID 11192870